CLINICAL TRIAL: NCT00120770
Title: Randomized Controlled Trial of Cellulose Sulfate Gel and HIV in Nigeria
Brief Title: Cellulose Sulfate (CS) Gel and HIV in Nigeria
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was halted in January 2007 due to safety concerns.
Sponsor: FHI 360 (Other)
Collaborators: Lagos State University (Other); University of Port Harcourt Teaching Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 9757
Record Dates: First submitted 2005-07-11; First posted 2005-07-19 (Estimated); Last update posted 2007-02-28 (Estimated); Status verified 2007-02

CONDITIONS: HIV Infections; Gonorrhea; Chlamydia Infections
Keywords: AE adverse event; AIDS acquired immunodeficiency syndrome; ALT (SGPT) alanine aminotransferase; ART antiretroviral therapy; AST (SGOT) aspartate aminotransferase; DCF data collection forms; DMC Data Monitoring Committee; FDA (U.S.) Food and Drug Administration; GCP Good Clinical Practice guidelines; HB sAg Hepatitis B surface antigen; ICH International Conference of Harmonisation; IND Investigational New Drug Application; IRB Institutional Review Board; IU international units; mg milligram(s); mm3 cubic millimeter(s); PCR polymerase chain reaction; SAE serious adverse event; µg microgram; ULN upper limit of the normal range; WB Western Blot; Human Immunodeficiency Virus; Neisseria gonorrhoeae; Chlamydia trachomatis; HIV Seronegativity
MeSH Terms: conditions — HIV Infections; Gonorrhea; Chlamydia Infections; Acquired Immunodeficiency Syndrome | interventions — Anti-Infective Agents

INTERVENTIONS:
Drug: Cellulose Sulfate Vaginal Gel (Microbicide)

SUMMARY:
This is a Phase 3, multi-center, randomized, placebo-controlled trial to determine the effectiveness and safety of the 6% cellulose sulfate (CS) vaginal gel for the prevention of HIV infection.

DETAILED DESCRIPTION:
This is a Phase 3, multi-center, randomized, placebo-controlled trial to assess the effectiveness of CS gel in preventing male-to-female vaginal transmission of HIV among HIV sero-negative women at high risk for HIV infection. Eligible participants who are HIV negative, at risk for becoming infected, and are willing to use a vaginal microbicide each time they have intercourse throughout 12 months of study participation will be recruited in Port Harcourt and Lagos, Nigeria. The enrollment phase will last until 2,160 women have enrolled. It is anticipated that the enrollment will be completed within 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give informed consent
* At least 18 years old and not more than 35 years old
* Average of three vaginal coital acts per week with a male partner
* More than one male sexual partner in the last 3 months
* Willing to use study product as directed
* Willing to adhere to follow-up schedule
* Willing to participate in the study for 12 months
* Willing to report self-medication during study participation
* Willing to give urine for pregnancy testing; self-administered vaginal swabs for GC/CT testing; OMT for HIV monthly; finger prick for HIV confirmation if required; and blood draw for syphilis and HIV at baseline, and for HIV at the final visit
* Willing to not use a spermicide, other vaginal contraceptive, or vaginal lubricant during the study
* At least 3 months since end of the last pregnancy

Exclusion Criteria:

* History of adverse reactions to the study products, including latex
* Pregnant or desire a pregnancy during the 12 months of participation
* Injection drug user
* Gynecological abnormality that may have an impact on the safety and/or response to the study gel according to the investigator
* HIV positive as diagnosed by OraQuick® rapid test
* Participation in any other microbicide research
* Discontinued from the CS study previously
* Any condition (social or medical) which, in the opinion of the investigator, would make study participation unsafe or complicate data interpretation

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2160
Dates: Start 2004-11; Study Completion 2007-03

PRIMARY OUTCOMES:
Incidence of HIV-1 and HIV-2 infection as determined by detection of HIV antibodies from oral mucosal transudate (OMT) specimens.

SECONDARY OUTCOMES:
Incidence of genital gonorrhea or chlamydia as determined by DNA probe technology from self-administered vaginal swabs.

CONTACTS AND LOCATIONS:
Overall Officials: Vera Halpern, MD, Study Director — FHI 360
Locations (2):
- Nigeria (2):
  - Lagos University, College of Medicine, Center 10151, Lagos
  - University of Port Harcourt Teaching Hospital, Center 10152, Port Harcourt

REFERENCES:
- [Derived] Halpern V, Obunge O, Ogunsola F, Otusanya S, Umo-Otong J, Wang CH, Mehta N. Interim data monitoring to enroll higher-risk participants in HIV prevention trials. BMC Med Res Methodol. 2009 Jun 23;9:44. doi: 10.1186/1471-2288-9-44. PMID 19549331
- [Derived] Halpern V, Ogunsola F, Obunge O, Wang CH, Onyejepu N, Oduyebo O, Taylor D, McNeil L, Mehta N, Umo-Otong J, Otusanya S, Crucitti T, Abdellati S. Effectiveness of cellulose sulfate vaginal gel for the prevention of HIV infection: results of a Phase III trial in Nigeria. PLoS One. 2008;3(11):e3784. doi: 10.1371/journal.pone.0003784. Epub 2008 Nov 21. PMID 19023429
- See also: Related Info — http://www.fhi.org
- See also: Related Info — http://conrad.org